CLINICAL TRIAL: NCT05494541
Title: Characteristics of Patients With Sickle Cell Disease Who Initiate Crizanlizumab Therapy
Brief Title: Characteristics of Patients With Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CSEG101AUS17
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Sickle Cell Disease
Keywords: Crizanlizumab,; sickle cell disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — crizanlizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Overall cohort: All the patients who met the base inclusion criteria were included in the cohort.
  Interventions: Other: Crizanlizumab
- Three-month cohort (3m cohort): Patients with stability and eligibility in IQVIA Patient Centric Medical Claims Database (Dx) and stability and eligibility in IQVIA Longitudinal Prescription Database (LRx) during the 3 months following the index date were included in the cohort.
  Interventions: Other: Crizanlizumab
- Six-month cohort (6m cohort): A subset of patients from the 3m cohort with stability and eligibility in Dx and stability and eligibility in LRx during the 6 months following the index date were included in this cohort.
  Interventions: Other: Crizanlizumab

INTERVENTIONS:
Other: Crizanlizumab — Patients who initiated crizanlizumab between November 1, 2019 and January 31, 2021 (index period) were selected into the treatment cohort.

SUMMARY:
This was a retrospective descriptive analysis of health care claims data using the IQVIA open source medical and pharmacy claims databases.

DETAILED DESCRIPTION:
Patients with a diagnosis of SCD between November 1, 2018 and April 30, 2021 were identified. Among these patients, those who initiated crizanlizumab between November 1, 2019 and January 31, 2021 (index period) were selected into the treatment cohort. The indexing timeframe allowed for a 1-year lookback period and a minimum of 3 months (3m cohort) of follow-up. A subset of the 3m cohort with 6-months of available (6m cohort) follow-up was performed. The index date was the date of the first crizanlizumab administration.

Study period: 01 November 2018 - 30 April 2021 Index period: 01 November 2019 - 31 January 2021 Index date: Date of the first claim for administration of crizanlizumab in the index period

ELIGIBILITY:
Inclusion Criteria:

* At least 1 claim in IQVIA Patient Centric Medical Claims Database (Dx) with SCD diagnosis (ICD-10 D57.xx, except D57.3) within the study period;
* At least 1 claim for administration of crizanlizumab within the index period. Index date was the date of first administration;
* At least 1 claim with HCPCs for crizanlizumab (J0791) OR with at least one claim for an unspecified biologic (J3590) on the same day as a claim for SCD (ICD-10 D57.xx, except D57.3) OR with at least one claim with HCPCs C9053;
* At least 16 years of age on the index date;
* Linkage to the IQVIA Longitudinal Prescription Database (LRx) within the study period;
* Stability and eligibility in Dx during the 12 months prior to the index date;
* Stability and eligibility in LRx during the 12 months prior to the index date

Exclusion Criteria:

* None

Ages: 16 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study included patients with SCD who initiated crizanlizumab in a real-world setting
Sampling Method: Non-Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-10-27 (Actual); Study Completion 2021-10-27 (Actual)

PRIMARY OUTCOMES:
Age | Baseline
  Age information was reported.
Number of patients: Gender | Baseline
  Gender information was reported.
Number of patients: Geographic region | Baseline
  The following categories were included:
  Northeast, Midwest, South, West
Number of patients: Insurance type | Baseline
  When multiple payer types were observed, the following hierarchy was used: Medicare, Commercial, Medicaid, Cash, Unspecifed.
  When commercially-managed Medicaid was observed, the Medicaid designation was assigned.
Number of patients by Charlson Comorbidity Index (CCI) score category | Baseline
  Severity of comorbidity was categorized into three grades: mild, with CCI scores of 1-2; moderate, with CCI scores of 3-4; and severe, with CCI scores ≥5.
Number of patients by comorbidity | Baseline
  Number of patients by IQVIA's standard comorbidity list were reported.
Number of patients with history of additional SCD-related comorbidities associated with organ damage | Baseline
  Number of patients with history of additional SCD-related comorbidities associated with organ damage were reported.
Number of patients : History of hydroxyurea use | Baseline
  Pre-index treatment history for sickle cell disease was reported.
Number of patients : History of L-glutamine use | Baseline
  Pre-index treatment history for sickle cell disease was reported.
Number of patients : History of Voxelotor use | Baseline
  Pre-index treatment history for sickle cell disease was reported.
Number of patients : SCD genotype | Baseline
  Number of patients with sickle cell disease genotype were reported.

SECONDARY OUTCOMES:
Proportion of patients with claims for hydroxyurea while on crizanlizumab therapy | Throughout the follow-up period, approximately 1.5 years
  Concomitant SCD treatments after initiating crizanlizumab
Number of hydroxyurea claims | Throughout the follow-up period, approximately 1.5 years
  Concomitant SCD treatments after initiating crizanlizumab
Proportion of patients with claims for L-glutamine while on crizanlizumab therapy | Throughout the follow-up period, approximately 1.5 years
  Concomitant SCD treatments after initiating crizanlizumab
Number of L-glutamine claims | Throughout the follow-up period, approximately 1.5 years
  Concomitant SCD treatments after initiating crizanlizumab
Proportion of patients with claims for voxelotor while on crizanlizumab therapy | Throughout the follow-up period, approximately 1.5 years
  Concomitant SCD treatments after initiating crizanlizumab
Number of voxelotor claims | Throughout the follow-up period, approximately 1.5 years
  Concomitant SCD treatments after initiating crizanlizumab

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CSEG101AUS17 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17968